CLINICAL TRIAL: NCT05430217
Title: Double-blind Placebo-controlled Multicenter Randomized Clinical Trial to Evaluate the Efficacy and Safety of Buspirone, Sustained-release Tablets, 15 mg (JSC Valenta Pharm, Russia) in Patients With Autonomic Dysfunction Syndrome Accompanied by Vertigo
Brief Title: Efficacy and Safety of Buspirone, Sustained-release Tablets, 15 mg in Patients With Autonomic Dysfunction Syndrome Accompanied by Vertigo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valenta Pharm JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BUSP-03-03-2021
Record Dates: First submitted 2022-06-14; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Vertigo; Autonomic Dysfunction
MeSH Terms: conditions — Vertigo; Primary Dysautonomias | interventions — Buspirone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buspirone, sustained-release tablets, 15 mg (Experimental): 15 mg/day
  Interventions: Drug: Buspirone
- Placebo (Placebo Comparator): 1 placebo tablet/day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Buspirone — 1 tablet (15 mg) once per day for 28 days
  Arms: Buspirone, sustained-release tablets, 15 mg
Drug: Placebo — 1 placebo tablet once per day for 28 days
  Arms: Placebo

SUMMARY:
Study to evaluate the efficacy and safety of Buspirone, sustained-release tablets, 15 mg in patients with autonomic dysfunction syndrome accompanied by vertigo

ELIGIBILITY:
Inclusion Criteria:

1. Signing and dating the patient's Informed Consent Form.
2. Women and men between the ages of 18 and 65, inclusive, at the time of signing the Informed Consent Form.
3. Clinical diagnosis: G90.8 Other autonomic nervous system disorders or G90.9 Autonomic nervous system disorder not specified.
4. Presence of dizziness, total DHI score from 36 to 52 points inclusive.
5. For women of preserved reproductive potential, a negative pregnancy test and agreement to use approved contraceptive methods for the duration of study participation, beginning at visit 0, and for 3 weeks after study termination; for men, agreement to use approved contraceptive methods for the duration of study participation and for 3 weeks after study termination.

Allowed contraceptive methods in this study are: intrauterine device, barrier method, or dual barrier method (condom or occlusion cap (diaphragm or cervical/vaulted cap) plus spermicide). Hormonal contraception is not permitted due to insufficient data on drug interactions of buspirone.

Women with infertility (menopausal (defined as not menstruating for at least 2 years or more) or with documented surgical sterilization (hysterectomy, bilateral oophorectomy, fallopian tubal ligation) and men with documented infertility or vasectomy are also eligible for participation.

Exclusion Criteria:

1. Known or suspected hypersensitivity to the active ingredient or any of the excipients of the study drug/placebo.
2. Lactose intolerance, lactase deficiency, glucose-galactose malabsorption.
3. Cumulative score > 2 on the Suicide Risk Assessment Scale.
4. Cumulative score > 16 on the Hamilton Scale.
5. Chronic heart failure New York Heart Association (NYHA) functional class III-IV, angina III-IV.
6. Syncopal and presyncopal conditions, including a history.
7. Acute cardiovascular disease or surgery (myocardial infarction, angioplasty, aortocoronary/mammary coronary artery bypass surgery, unstable angina, etc) less than 6 months before the screening visit.
8. Acute cerebral circulation disorders and/or transient ischemic attacks less than 6 months before the screening visit date.
9. Cardiac rhythm and conduction disorders, including a history. An established artificial pacemaker.
10. Established diagnosis of liver failure, including a history and/or changes in liver enzyme activity:

    * increased aspartate aminotransferase (AST), alanine aminotransferase (ALT) more than 2.5 times the upper limit of normal,
    * increase in the level of total bilirubin more than 1.5 times above the upper limit of normal;
    * Prothrombin time >18 s.

Chronic kidney disease history of stage IIIa-V (as defined by the National Kidney Foundation/Kidney Disease Outcomes Quality Initiative, NKF/KDOQI, 2006).

12. Glomerular filtration rate (GFR) ≤ 60 mL/min, calculated using the CKD-EPI equation, based on serum creatinine levels at screening.

13. Diabetes mellitus of moderate and severe severity, as well as mild subcompensation and decompensation.

14. Myasthenia gravis. 15. Glaucoma. 16. Systemic connective tissue diseases. 17. Autoimmune diseases. 18. The need for surgical and/or endovascular treatment in the next 3 months. 19. Epilepsy or seizures of unclear etiology, including a history of seizures. 20. Alcoholism, drug addiction, substance abuse in the history and/or at the time of screening (alcoholism - use of more than 30 ml of ethyl alcohol per day within the last 6 months; drug addiction - use of any narcotic substances in any dose within the last 6 months; substance abuse - use of any psychoactive substances in any dose within the last 6 months).

21. Schizophrenia, schizoaffective disorder, history of bipolar disorder. 22. Tuberculosis, hepatitis B and C, HIV, syphilis, history or screening results.

23. Conditions after surgical operations, if less than 6 months have passed since the operation.

24. Therapy for cognitive impairment, balance disorders, and dizziness 21 days or less before the date of Visit 1.

25. Use of an irreversible MAO inhibitor within 14 days or a reversible MAO inhibitor within 1 day before Visit 1.

26. Therapy with the following drugs and groups of drugs: 7 days or less before screening:

* Selective serotonin reuptake inhibitors (SSRIs) and selective serotonin and noradrenaline reuptake inhibitors (SSNs);
* Betahistine preparations;
* Cytochrome P450 3A4 (CYP3A4) inhibitors and inducers: erythromycin, itraconazole, nefazodone, diltiazem, verapamil, etc;
* Cimetidine, warfarin, phenytoin, propranolol.

Monoamine oxidase inhibitors (MAOIs):

Do not use MAO inhibitors concomitantly or take the drug earlier than 14 days after withdrawal of an irreversible MAO inhibitor, or less than 1 day after withdrawal of a reversible MAO inhibitor.

27. History of malignancy, except for patients who have not had the disease within the last 5 years, patients with fully cured basal cell carcinoma of the skin, or fully cured carcinoma in situ.

28. Decompensated somatic diseases that, in the opinion of the investigator, would prevent the patient from following the regimen prescribed by the study protocol, or would not allow evaluation of therapy and compliance in accordance with the protocol, or could distort the results of the study.

29. Decompensated neuropsychiatric conditions, including multiple sclerosis, Parkinson's disease, endogenous depression or other conditions that, in the opinion of the investigator, will not permit the patient to follow the regimen prescribed by the research protocol or will not permit an evaluation of treatment effectiveness and compliance in accordance with the protocol, or may skew the results of the study.

30. Women who are pregnant or lactating; women planning to become pregnant within the next 2 months.

31. Patient using or planning to use hormonal contraception during the study 32. Patients who need concomitant therapy prohibited in this study. 33. Participation in another clinical trial within the last 3 months prior to the screening visit date.

34. Acute intoxication caused by alcohol, sleeping pills, analgesics, antipsychotics.

35. Patient's unwillingness or inability to comply with protocol procedures (in the opinion of the study physician).

36. Other conditions that, in the opinion of the Researcher, prevent the patient from being included in the study.

37. Patient is diagnosed with COVID-19 disease at the time of screening; or has symptoms of SARS or COVID-19 within 14 days prior to screening and has a positive rapid test for COVID-19 at screening.

Withdrawal Criteria:

1. Patient's desire to stop participating in the study.
2. Researcher's decision that continued participation in the study is contrary to the patient's best interests.
3. Patient's inclusion in the study in violation of the inclusion and non-inclusion criteria.
4. Researcher's decision to exclude the patient from the study because the patient did not cooperate adequately with the researcher during the study.
5. Skipping 3 or more consecutive study drug/placebo tablets or skipping 6 or more study drug/placebo tablets.
6. Unwanted event requiring withdrawal of study therapy or limiting protocol procedures.
7. Need to prescribe a patient medication from the Prohibited Companion Therapies section.
8. Loss of communication with the patient.
9. Pregnancy of the patient.
10. For each research visit: patient diagnosed with COVID-19 disease at the time of the visit; or presence of symptoms of ARI or COVID-19 within 7 days prior to the research visit and a positive rapid test for COVID-19 at the research visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2022-01-28 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-05-09 (Actual)

PRIMARY OUTCOMES:
Frequency of response to therapy at Visit 5 | Visit 5 (day 28±1)
  A number (%) of patients with reduction of ≥50% in the total Dizziness Handicap Inventory (DHI) score (25-item self-report questionnaire with total score from 0 to 100; higher scores mean a worse outcome) compared to Visit 1

SECONDARY OUTCOMES:
Frequency of response to therapy at Visits 2, 3, and 4. | Visit 2 (day 7±1), Visit 3 (day 14±1), Visit 4 (day 21±1)
  A number (%) of patients with reduction of ≥50% in the total Dizziness Handicap Inventory (DHI) score (25-item self-report questionnaire with total score from 0 to 100; higher scores mean a worse outcome) compared to Visit 1
Total score on the DHI Scale at Visits 2, 3, 4, and 5. | Visit 2 (day 7±1), Visit 3 (day 14±1), Visit 4 (day 21±1), Visit 5 (day 28±1)
  Total Dizziness Handicap Inventory (DHI) score (25-item self-report questionnaire with total score from 0 to 100; higher scores mean a worse outcome)
Change in total DHI score on Visits 2, 3, 4, and 5 compared to Visit 1 | Visit 2 (day 7±1), Visit 3 (day 14±1), Visit 4 (day 21±1), Visit 5 (day 28±1)
  The difference between the total Dizziness Handicap Inventory (DHI) score (25-item self-report questionnaire with total score from 0 to 100; higher scores mean a worse outcome) on Visit 2-5 and Visit 1
Proportion of patients with a 30% or greater reduction in DHI score compared to baseline by Visit 2, 3, 4, 5 | Visit 2 (day 7±1), Visit 3 (day 14±1), Visit 4 (day 21±1), Visit 5 (day 28±1)
  A number (%) of patients with reduction of ≥30% in the total Dizziness Handicap Inventory (DHI) score (25-item self-report questionnaire with total score from 0 to 100; higher scores mean a worse outcome) compared to Visit 1
Time elapsed before the total DHI score decreased by 50% or more from baseline | Day 1 - Day 28±1
  Time (days) elapsed before a ≥50% decrease in Dizziness Handicap Inventory (DHI) score (25-item self-report questionnaire with total score from 0 to 100; higher scores mean a worse outcome)
Time elapsed before the total DHI score decreased by 30% or more from baseline | Day 1 - Day 28±1
  Time (days) elapsed before a ≥30% decrease in Dizziness Handicap Inventory (DHI) score (25-item self-report questionnaire with total score from 0 to 100; higher scores mean a worse outcome)
Change in digital rating scale (DRS) score from Visit 1 to Visits 2, 3, 4, 5 | Visit 2 (day 7±1), Visit 3 (day 14±1), Visit 4 (day 21±1), Visit 5 (day 28±1)
  The difference between the total DRS score (from minimum of 0 to maximum of 10 points; higher scores mean a worse outcome) on Visit 2-5 and Visit 1
Ddigital rating scale (DRS) score on Visit 2, 3, 4, and 5 | Visit 2 (day 7±1), Visit 3 (day 14±1), Visit 4 (day 21±1), Visit 5 (day 28±1)
  DRS score (from minimum of 0 to maximum of 10 points; higher scores mean a worse outcome) on the Visit
The response on the Likert scale at Visits 2, 3, 4, and 5 | Visit 2 (day 7±1), Visit 3 (day 14±1), Visit 4 (day 21±1), Visit 5 (day 28±1)
  Percentage of patients with complete response, significant relief, moderate relief, minor relief, and no response on the Likert scale at Visits 2, 3, 4, and 5.

OTHER OUTCOMES:
Safety and Tolerability: adverse event (AE) number and frequency | From the screening to Visit 6 (day 35±1)
  Number and frequency of adverse events (AEs)
Safety and Tolerability: serious AEs (SAEs) number and frequency | From the screening to Visit 6 (day 35±1)
  Number and frequency of serious AEs (SAEs)
Safety and Tolerability: AE and SAE causal relationship | From the screening to Visit 6 (day 35±1)
  Number and frequency of AEs and SAEs related to the use of the study drug/placebo
Safety and Tolerability: Percentage of patients who interrupted treatment due to AE | From the screening to Visit 6 (day 35±1)
  Number and percentage of patients who interrupted treatment due to AE
Safety and Tolerability: vital signs - systolic blood pressure (SBP) | From the screening to Visit 6 (day 35±1)
  SBP, mmHg
Safety and Tolerability: vital signs - diastolic blood pressure (DBP) | From the screening to Visit 6 (day 35±1)
  DBP, mmHg
Safety and Tolerability: vital signs - respiratory rate (RR) | From the screening to Visit 6 (day 35±1)
  RR, breaths per minute
Safety and Tolerability: vital signs - heart rate (HR) | From the screening to Visit 6 (day 35±1)
  HR, beats per minute
Safety and Tolerability: vital signs - body temperature | From the screening to Visit 6 (day 35±1)
  Body temperature, centigrade scale
Safety and Tolerability: physical examination results | From the screening to Visit 6 (day 35±1)
  Any patient complaints or abnormalities found during examination by a general practitioner
Safety and Tolerability: results of the neurological examination | From the screening to Visit 6 (day 35±1)
  Any patient complaints or abnormalities found during examination by a neurologist
Safety and Tolerability: complete blood count - hemoglobin | From the screening to Visit 6 (day 35±1)
  Hemoglobin, g/dL
Safety and Tolerability: complete blood count - hematocrit | From the screening to Visit 6 (day 35±1)
  Hematocrit, %
Safety and Tolerability: complete blood count - red blood cells | From the screening to Visit 6 (day 35±1)
  Red blood cells, 10^6/uL
Safety and Tolerability: complete blood count - white blood cells | From the screening to Visit 6 (day 35±1)
  White blood cells, 10^3/uL
Safety and Tolerability: complete blood count - neutrophils | From the screening to Visit 6 (day 35±1)
  Neutrophils, %
Safety and Tolerability: complete blood count - lymphocytes | From the screening to Visit 6 (day 35±1)
  Lymphocytes, %
Safety and Tolerability: complete blood count - eosinophils | From the screening to Visit 6 (day 35±1)
  Eosinophils, %
Safety and Tolerability: complete blood count - Monocytes | From the screening to Visit 6 (day 35±1)
  Monocytes, %
Safety and Tolerability: complete blood count - basophils | From the screening to Visit 6 (day 35±1)
  Basophils, %
Safety and Tolerability: complete blood count - platelets | From the screening to Visit 6 (day 35±1)
  Platelets, 10^3/uL
Safety and Tolerability: complete blood count - erythrocyte sedimentation rate | From the screening to Visit 6 (day 35±1)
  Erythrocyte sedimentation rate, mm per hour
Safety and Tolerability: blood test results - alanine transaminase (ALT) | From the screening to Visit 6 (day 35±1)
  ALT in blood serum, U/L
Safety and Tolerability: blood test results - aspartate transaminase (AST) | From the screening to Visit 6 (day 35±1)
  AST in blood serum, U/L
Safety and Tolerability: blood test results - total bilirubin | From the screening to Visit 6 (day 35±1)
  Total bilirubin in blood serum, umol/L
Safety and Tolerability: blood test results - glucose | From the screening to Visit 6 (day 35±1)
  Glucose in blood serum, mmol/L
Safety and Tolerability: blood test results - total protein | From the screening to Visit 6 (day 35±1)
  Total protein in blood serum, g/L
Safety and Tolerability: blood test results - creatinine | From the screening to Visit 6 (day 35±1)
  Creatinine in blood serum, umol/L
Safety and Tolerability: blood test results - urea | From the screening to Visit 6 (day 35±1)
  Urea in blood serum, mmol/L
Safety and Tolerability: blood test results - prothrombin time | From the screening to Visit 6 (day 35±1)
  Prothrombin time, s
Safety and Tolerability: urinalysis - pH | From the screening to Visit 6 (day 35±1)
  pH of the urine
Safety and Tolerability: urinalysis - specific gravity | From the screening to Visit 6 (day 35±1)
  Specific gravity of the urine
Safety and Tolerability: urinalysis - glucose | From the screening to Visit 6 (day 35±1)
  Glucose in the urine (mmol/L)
Safety and Tolerability: urinalysis - protein | From the screening to Visit 6 (day 35±1)
  Protein in the urine (g/L)
Safety and Tolerability: urinalysis (microscopy) - red blood cells | From the screening to Visit 6 (day 35±1)
  Red blood cells in the urine (number in sight)
Safety and Tolerability: urinalysis (microscopy) - white blood cells | From the screening to Visit 6 (day 35±1)
  White blood cells in the urine (number in sight)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - heart rate | From the screening to Visit 6 (day 35±1)
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: heart rate (beats per minute)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - PQ interval | From the screening to Visit 6 (day 35±1)
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: PQ interval (ms)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - QRS complex | From the screening to Visit 6 (day 35±1)
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: QRS complex (ms)
Safety and Tolerability: 12-lead electrocardiogram (ECG) - corrected QT interval (QTc) | From the screening to Visit 6 (day 35±1)
  12-lead ECG (I, II, III, aVR, aVL, aVF, V1-V6) taken while lying down: QTc (ms)
Exploratory: total score on the Hamilton scale | Visit 4 (day 21±1), Visit 5 (day 28±1)
  Total score on the Hamilton scale (21-item scale with total score from 0 to 52; higher scores mean a worse outcome)
Exploratory: change in total score on the Hamilton scale compared to Visit 1 | Visit 4 (day 21±1), Visit 5 (day 28±1)
  Difference between the score on the Hamilton scale (21-item scale with total score from 0 to 52; higher scores mean a worse outcome) on Visit 4 or 5 and Visit 1

CONTACTS AND LOCATIONS:
Locations (8):
- Russia (8):
  - Regional budgetary health care institution "Ivanovo Regional Clinical Hospital", Saint Petersburg
  - Limited Liability Company "Research Center Eco-Security", Saint Petersburg
  - Limited Liability Company "X7 Clinical Research", Saint Petersburg
  - Limited Liability Company "Research Center Eco-Safety", Saint Petersburg
  - Limited Liability Company "MK-Med", Saint Petersburg
  - Saint Petersburg State Budgetary Institution of Healthcare "City Hospital No. 40 of Kurortny District", Saint Petersburg
  - St. Petersburg State Budgetary Health Institution "City Polyclinic No. 106", Saint Petersburg
  - Limited Liability Company "MART", Saint Petersburg

IPD SHARING:
Plan to Share IPD: Undecided